CLINICAL TRIAL: NCT04227561
Title: Analgesia for Pediatric Circumcision : Comparison of the Effectiveness of Neurostimulation-guided Pudendal Nerve Block to Ultrasound-guided Penile Nerve Block
Brief Title: Analgesia for Pediatric Circumcision : Comparison of the Effectiveness of Pudendal Nerve Block to Penile Nerve Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B076201941947
Record Dates: First submitted 2019-12-20; First posted 2020-01-13 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Anesthesia; Pediatric Circumcision
Keywords: penile nerve block; pudendal nerve block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pudendal nerve block (Active Comparator): Neurostimulation-guided pudendal nerve block
  Interventions: Procedure: Pudendal nerve block
- Penile nerve block (Active Comparator): Ultrasound-guided penile nerve block
  Interventions: Procedure: Penile nerve block

INTERVENTIONS:
Procedure: Pudendal nerve block — Pudendal nerve block will be performed under general anesthesia and guided by neurostimulation.
  The local anesthetic solution (chirocaine 2.5mg/ml) will be injected in the ischiorectal fossa with a needle (a BBraun Stimuplex Ultra 360 22G 50mm needle) connected to a neurostimulator (Stimuplex HNS 12 neurostimulator). The neurostimulator will be used to determine the localization of pudendal nerve and to identify the precise site of injection. The contraction of the anal sphincter or bulbocavernosus muscle occurs when the pudendal nerve is reached.
  These procedure will be performed bilaterally.
  Arms: Pudendal nerve block
Procedure: Penile nerve block — The local anesthetic solution (chirocaine 2.5mg/ml) will be injected under the fascia of Scarpa with a real-time ultrasound guidance.
  These procedure will be performed bilaterally.
  Arms: Penile nerve block

SUMMARY:
Medical or ritual circumcisions are frequent interventions in children. To provide the best comfort to the patients, the anesthetists use regional anesthesia. Complementary to general anesthesia, this method allows to lower the need of opioids during and after the surgery, as well as a faster recovery.

The foreskin is innervated by the dorsal nerve of the penis which is the branch of the pudendal nerve. This nerve arises from the sacral plexus and more precisely the branches S2-3-4. There are two methods to block pudendal nerve. First, the pudendal nerve block is an old anesthetic technique developed in 1908, first for obstetrical analgesia and urological analgesia. It consists in injecting in the ischiorectal fossa, right at the end of Alcock's canal, a solution of local anesthetic. Second, the penile nerve block, described in the middle of the seventies, consists in injecting a solution of local anesthetic that blocks only the terminal part of the pudendal nerve.

Those two nerve blocks have been subject to many publications, especially concerning the method to apply to optimize their efficiency. The literature review led to this conclusion: The penile nerve block should be ultrasound guided and the pudendal nerve block should be done with a neurostimulator.

The aim of this study is to compare the analgesic efficiency of the ultra-sound guided penile nerve block to the pudendal nerve block with neurostimulation, for the pediatric circumcision.

ELIGIBILITY:
Inclusion Criteria:

* One to two years old boys
* Ritual or medical, elective circumcision.

Exclusion Criteria:

* Refusal from parents
* Allergy to local anesthetics
* Documented coagulation disorders
* Epilepsy

Ages: 1 Year to 2 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2020-01-17 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Time to first administration of analgesics (other than nervous blockage after induction of anesthesia) | up to 24 hours
  Pain evaluation during surgery will be based on hemodynamic fluctuations (elevation of 15% or more of the heart rate or blood pressure) and variations of skin conductance (Med-Storm's pain monitor). In the postoperative period, the pain will be evaluated with the EVENDOL score and the variations of skin conductance

SECONDARY OUTCOMES:
Postoperative pain assessed with the EVENDOL score | up to 24 hours
  Pain will be assessed with the EVENDOL score (score 0 to 15) at T0 (upon arrival in the recovery room), T1 (30 minutes post-surgery), T2 (1 hour post-surgery), T3 (3 hours post-surgery). EVENDOL scale is a behavioral pain scale for children aged 0 to 7 years.
Postoperative pain assessed by a pain monitor device (skin conductance algesimeter) | up to 24 hours
  Continuous variations of skin conductance will be measured and analyzed during the operation

CONTACTS AND LOCATIONS:
Overall Officials: Panayota Kapessidou, MD,PhD, Study Director — University Hospital Saint-Pierre (CHU Saint-Pierre), Université Libre de Bruxelles (ULB); Alexandros Alexis, MD, Principal Investigator — University Hospital Saint-Pierre (CHU Saint-Pierre), Université Libre de Bruxelles (ULB); Olivier Habchi, MD, Principal Investigator — University Hospital Saint-Pierre (CHU Saint-Pierre), Université Libre de Bruxelles (ULB)
Locations (1):
- University Hospital Saint-Pierre, Université Libre de Bruxelles (ULB), Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faraoni D, Gilbeau A, Lingier P, Barvais L, Engelman E, Hennart D. Does ultrasound guidance improve the efficacy of dorsal penile nerve block in children? Paediatr Anaesth. 2010 Oct;20(10):931-6. doi: 10.1111/j.1460-9592.2010.03405.x. PMID 20849498
- [Background] Sandeman DJ, Dilley AV. Ultrasound guided dorsal penile nerve block in children. Anaesth Intensive Care. 2007 Apr;35(2):266-9. doi: 10.1177/0310057X0703500217. PMID 17444318
- [Background] Gjerstad AC, Wagner K, Henrichsen T, Storm H. Skin conductance versus the modified COMFORT sedation score as a measure of discomfort in artificially ventilated children. Pediatrics. 2008 Oct;122(4):e848-53. doi: 10.1542/peds.2007-2545. PMID 18829782
- [Background] Bateman DV. An alternative block for the relief of pain of circumcision. Anaesthesia; 1975, 30:101-2
- [Background] Müller B. Narkologie. Band II, 88. Berlin: Trankel; 1908. p.15.
- [Background] B. Dalens. Traité d'anesthésie générale. Arnette,11/01. ISBN: 2-7184-1022-1.